CLINICAL TRIAL: NCT01661140
Title: Randomized, Phase IV, Placebo-controlled, Comparative Study to Evaluate the Efficacy and Safety of Tapering Methotrexate (MTX) Dosage Versus Maintaining the Dosage in Patients With Severe Active Rheumatoid Arthritis (RA) Who Have Demonstrated an Inadequate Response (IR) to Prior Disease-modifying Anti-rheumatic Drugs (DMARDs) Treatment and Have Initiated RoActemra (RoActemra, TCZ) in Combination With MTX
Brief Title: A Study of RoActemra/Actemra (Tocilizumab) in Combination With Methotrexate in Patients With Severe Active Rheumatoid Arthritis, Comparing Tapering Versus Maintaining the Methotrexate Dosage
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML28096; 2011-005260-20 (EudraCT Number)
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Results first posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; tocilizumab; Drug Tapering

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Methotrexate (MTX) Tapering Dosage (Experimental): At Week 0 participants will start open-label tocilizumab and open-label MTX for 24 weeks. At Week 24, participants achieving a good/moderate European League Against Rheumatism (EULAR) disease response will be randomized to the MTX Tapering group or MTX Maintenance group. In this arm participants will receive a double-blind MTX dose according to the MTX tapering scheme between Week 24 and Week 56. Participants will also continue to receive open-label tocilizumab between Week 24 and Week 56. From Week 56 to Week 72 participants will receive tocilizumab monotherapy.
  Interventions: Drug: Tocilizumab; Drug: Methotrexate (tapering dose)
- Methotrexate (MTX) Maintenance Dosage (Active Comparator): At Week 0 participants will start open-label tocilizumab and open-label MTX for 24 weeks. At Week 24, participants achieving a good/moderate European League Against Rheumatism (EULAR) disease response will be randomized to the MTX Tapering group or MTX Maintenance group. In this arm participants will continue to be administered a stable dose of MTX in a double-blind fashion between Week 24 and Week 56. Participants will also continue to receive open-label tocilizumab between Week 24 and Week 56. From Week 56 to Week 72 participants will receive tocilizumab monotherapy.
  Interventions: Drug: Methotrexate (stable dose); Drug: Tocilizumab

INTERVENTIONS:
Drug: Methotrexate (stable dose) — Methotrexate (MTX) was administered weekly according to the subject's pre-study MTX dose
  Arms: Methotrexate (MTX) Maintenance Dosage
Drug: Tocilizumab — 8 mg/kg intravenously every 4 weeks for 72 weeks
  Other Names: RoActemra/Actemra
Drug: Methotrexate (tapering dose) — Tapering doses of methotrexate (MTX) were administered weekly from Week 24 to Week 56. Tapering doses depended on dose administered to the subject during the open label period. First tapering occurred at randomization (Week 24), second tapering at Week 32, third tapering at Week 40 and final tapering at Week 48.
  Arms: Methotrexate (MTX) Tapering Dosage

SUMMARY:
This randomized, placebo-controlled, double-blind study will compare the safety and efficacy of tapering methotrexate (MTX) versus maintaining MTX dosage in patients with severe active rheumatoid arthritis and an inadequate response to disease-modifying antirheumatic drugs (DMARDs) initiated on treatment with tocilizumab. Participants will receive tocilizumab 8 mg/kg intravenously every 4 weeks and MTX orally weekly throughout the study. At Week 24, participants achieving a good/moderate EULAR response will be randomized receiving the MTX Tapering arm or MTX Maintenance arm. Up to Week 56 participants will receive either tapering or stable dose MTX in combination with tocilizumab. From Week 56 to Week 72 participants will receive tocilizumab monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Active severe rheumatoid arthritis (DAS28 > 5.1) according to European League of Rheumatism (EULAR)/American College of Rheumatology (ACR) criteria
* Inadequate response to a trial of 2 DMARDs, including methotrexate, a trial being defined as 6 months with 2 months at standard dose; no previous treatment with a biologic agent such as a tumor necrosis factor (TNF) inhibitor
* Oral corticosteroids must have been at a stable dose of </= 10 mg/day prednisolone or equivalent for at least 25 out of 28 days prior to start of treatment (Day 1)

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization
* Rheumatic autoimmune disease other than rheumatoid arthritis
* Functional class IV as defined by the ACR Classification of Functional Status in RA
* Prior history of or current inflammatory joint disease other than RA
* Previous treatment with tocilizumab
* Previous treatment with any biologic drug (e.g. TNF inhibitor) that is used in the treatment of RA
* Intraarticular or parenteral corticosteroids within 6 weeks prior to enrollment
* Inadequate liver, bone marrow or hepatic function
* Positive for hepatitis B, hepatitis C or HIV infection
* Pregnant or breastfeeding women
* Females of child-bearing potential who are not using reliable means of contraception
* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies
* Active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections
* History of, or currently active, primary or secondary immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2012-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (63):
- United Kingdom (63):
  - Aberdeen
  - Abergavenny
  - Ashford
  - Aylesbury
  - Barnsley
  - Basingstoke
  - Bournemouth
  - Brighton
  - Bury Saint Edmonds
  - Cambridge
  - Cannock
  - Cardiff
  - Chelmsford
  - Chester
  - Coventry
  - Crewe
  - Darlington
  - Derby
  - Dudley
  - Dundee
  - Eastbourne
  - Exeter
  - Gillingham
  - Greenock
  - Guildford
  - Harrogate
  - Hull
  - Isle of Wight
  - Leeds
  - Liverpool
  - Llantrisant
  - London
  - Londonderry
  - Maidstone
  - Manchester
  - Metropolitan Borough of Wirral
  - Middlesbrough
  - North Shields
  - Northampton
  - Nottingham
  - Oldham
  - Plymouth
  - Reading
  - Salford
  - Salisbury
  - Sheffield
  - Somerset
  - Southampton
  - Southport
  - Stevenage
  - Stoke-on-Trent
  - Sunderland
  - Sutton in Ashfield
  - Swindon
  - Torquay
  - Truro
  - Walsall
  - Warwick
  - Westcliffe-on-sea
  - Wolverhampton
  - Worthing
  - Wrightington
  - York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The initial open label period of the study consisted of one group of 427 participants. After completion of the initial phase only participants, who achieved a good/moderate disease response, were randomized into the double blind period. 272 participants were randomized into the two arms entering the double-blind period of the study.
Groups:
- Initial Phase: At Week 0 participants started open-label tocilizumab and open-label methotrexate (MTX) for 24 weeks, which was the initial phase of the study.
- Methotrexate (MTX) Tapering Group: After the open-label period ended at Week 24, participants achieving a good/moderate European League Against Rheumatism (EULAR) disease response were randomized to the MTX Tapering Group or MTX Maintenance Group. In the MTX Tapering Group participants received a double-blind MTX dose according to the MTX tapering scheme between Week 24 and Week 56. In addition, participants continued to receive open-label tocilizumab between Week 24 and Week 56. From Week 56 to Week 72 participants received tocilizumab monotherapy.
- Methotrexate (MTX) Maintenance Group: After the open-label period ended at Week 24, participants achieving a good/moderate European League Against Rheumatism (EULAR) disease response were randomized to the MTX Tapering Group or MTX Maintenance Group. In the MTX Maintenance Group participants continued to be administered the same dose of MTX in a double-blind fashion from Week 25 to Week 56. In addition, participants continued to receive open-label tocilizumab from Week 25 to Week 56. From Week 56 to Week 72 participants received tocilizumab monotherapy.
Period: Open-Label Period
Arm/Group | Initial Phase | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Started | 427 (All participants entered the study in the initial phase for 24 weeks of open label treatment.) | 0 | 0
Completed | 351 | 0 | 0
Not Completed | 76 | 0 | 0
Not completed — Adverse Event | 44 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0
Not completed — Investigator Decision | 3 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Administrative/Other | 1 | 0 | 0
Not completed — Sponsor termination | 16 | 0 | 0
Not completed — Did not meet EULAR criteria | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Period: Double-Blind Period
Arm/Group | Initial Phase | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Started | 0 (Those with a good/moderate disease response in the initial phase were randomized to the MTX arms.) | 136 (Only those with a good/moderate disease response in the initial phase were randomized.) | 136 (Only those with a good/moderate disease response in the initial phase were randomized.)
Completed | 0 | 95 | 86
Not Completed | 0 | 41 | 50
Not completed — Refused Treatment | 0 | 0 | 1
Not completed — Adverse Event | 0 | 16 | 18
Not completed — Protocol Violation | 0 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 3
Not completed — Investigator's Decision | 0 | 1 | 2
Not completed — Sponsor Termination | 0 | 14 | 17
Not completed — Administrative/Other | 0 | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Initial Phase: At Week 0 participants started open-label tocilizumab and open-label MTX for 24 weeks.
Arm/Group | Initial Phase
Number analyzed (Participants) | 427
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 326
  Male | 101

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Previous Disease Activity (European League Against Rheumatism [EULAR] Response) From Week 24 (Time of Randomization) to Week 60
Description: Response was determined using EULAR criteria based upon (Disease Activity Score In 28 Joints) DAS28 absolute scores at the assessment visit and the DAS28 reduction from the reference visit. Participants with a score lesser than or equal to (<=) 3.2 and reduction of greater than (>) 1.2 points were assessed as having a 'good' response. Participants with a score >3.2 with reduction of >1.2 points, or a score <=5.1 with reduction of >0.6 to <=1.2 points, were assessed as having a 'moderate' response. Participants with a score >5.1 with reduction of >0.6 to <=1.2 points, or any score with reduction <=0.6 points, were assessed as non-responders with response recorded as 'none.'
Time Frame: From randomization to Week 60
Population: Intention to treat (ITT) population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 136 | 136
percentage of participants | 76.5 | 65.4
Statistical Analysis 1: Comparison: Methotrexate (MTX) Tapering Group vs Methotrexate (MTX) Maintenance Group; Comparison was Tapering MTX : MTX maintenance. Last post-baseline EULAR response recorded used for participants with a missing result at Week 60; Test type: Non-Inferiority or Equivalence — Non-inferiority if the difference between treatments is statistically significant and the lower limit of the 95% confidence interval (CI) is greater than 0.9; p = 0.036, Analysis by logistic regression; Odds Ratio (OR) = 1.803, 95% CI 2-sided [1.037 to 3.133]

2. Secondary Outcome: Change From Baseline in Disease Activity Score In 28 Joints (DAS28) Score at Week 60
Description: The DAS28 defined as a combined index for measuring disease activity in rheumatoid arthritis (RA). The index included swollen (range 0-28) and tender joint counts (TJC) (range 0-28), acute phase response Erythrocyte Sedimentation Rate (ESR), and general health status (range 1-100). The index was calculated using the following formula: The DAS28 was calculated as [0.28 x the square root of number of swollen joints] + [0.56 x the square root of number of tender joints] + [0.7 x the natural log of ESR] + [0.014 x patient global assessment of disease activity]. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity.
Time Frame: Randomization (Week 24), Week 60
Population: ITT population included all randomized participants. Here, number of participants analyzed signifies those participants who were evaluable for this end point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 136 | 136
units on a scale
  Baseline (n= 135, 136) | 2.572 (1.3218) | 2.573 (1.3017)
  Change at Week 60 (n= 134, 135) | -0.179 (1.1702) | -0.233 (1.5156)

3. Secondary Outcome: Change From Baseline in Disease Activity Score In 28 Joints (DAS28) Score at Week 72
Description: as for outcome 2
Time Frame: Randomization (Week 24), Week 72
Population: ITT population included all randomized participants. Here, number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 134 | 135
units on a scale | -0.105 (1.2262) | -0.224 (1.4961)

4. Secondary Outcome: Percentage of Participants Who Achieve Score of <=1 in Tender Joint Count (TJC) and Swollen Joint Count (SJC) at Week 60 and 72
Description: Percentage of participants who achieve score of =1 in TJC and SJC at week 60 and 72 were reported. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1; total was calculated by adding all the joints for a maximum score of 28. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1; total was calculated by adding all the joints for a maximum score of 28.
Time Frame: Week 60, 72
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 136 | 136
percentage of participants
  TJC <=1, Week 60 | 39.0 | 39.0
  SJC <=1, Week 60 | 44.1 | 58.1
  TJC <=1, Week 72 | 37.5 | 40.4
  SJC <=1, Week 72 | 55.9 | 60.3

5. Secondary Outcome: Percentage of Participants Who Achieve a Disease Activity Score In 28 Joints (DAS28) <= 3.2
Description: The DAS28 index was calculated using the following formula: The DAS28 was calculated as [0.28 x the square root of number of swollen joints] + [0.56 x the square root of number of tender joints] + [0.7 x the natural log of ESR] + [0.014 x patient global assessment of disease activity]. Participants who achieve score <=3.2 at weeks 60 and 72 were reported.
Time Frame: Week 60, 72
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 136 | 136
percentage of participants
  Week 60 | 59.6 | 62.5
  Week 72 | 61.0 | 60.3

6. Secondary Outcome: Percentage of Participants Who Achieve DAS28 Remission (DAS28 < 2.6)
Description: The DAS28 index was calculated using the following formula: The DAS28 was calculated as [0.28 x the square root of number of swollen joints] + [0.56 x the square root of number of tender joints] + [0.7 x the natural log of ESR] + [0.014 x patient global assessment of disease activity]. Participants who achieve DAS28 remission score <2.6 at weeks 60 and 72 were reported.
Time Frame: Week 60, 72
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 136 | 136
percentage of participants
  Week 60 | 51.5 | 47.1
  Week 72 | 50.0 | 51.5

7. Secondary Outcome: Percentage of Participants Who Achieve Change in Disease Activity Score (cDAS) >=1.2
Description: The DAS28 index was calculated using the following formula: The DAS28 was calculated as [0.28 x the square root of number of swollen joints] + [0.56 x the square root of number of tender joints] + [0.7 x the natural log of ESR] + [0.014 x patient global assessment of disease activity]. Participants who achieve cDAS28 >=1.2 score at weeks 60 and 72 were reported.
Time Frame: Week 60, 72
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 136 | 136
percentage of participants
  Week 60 | 9.6 | 16.2
  Week 72 | 9.6 | 15.4

8. Secondary Outcome: Percentage of Participants Who Achieve Clinical Disease Activity Index (CDAI) Remission (CDAI < 2.8) at Week 60 and 72
Description: Clinical Disease Activity Index (CDAI) was an index for measuring disease activity in RA. The index was calculated using the following formula: CDAI: SJC28 + TJC28 + patient global assessment of disease (PGA) 10 centimeter [cm] Visual Analog Scale [VAS] + physician global assessment of disease (PhGA) 10 cm VAS. VAS assessments involved a 10 cm horizontal scale from 'no disease activity' to 'maximum disease activity.' CDAI scores ranged from 0 to 76, with higher scores indicating increased disease activity.
Time Frame: Randomization (Week 24), Week 60, 72
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 136 | 136
percentage of participants
  Week 60 | 2.9 | 1.5
  Week 72 | 1.5 | 3.7

9. Secondary Outcome: Percentage of Participants Who Achieve Simplified Disease Activity Index (SDAI) Remission (SDAI < 3.3) at Week 60 and 72
Description: Simplified Disease Activity Index (SDAI) was an index for measuring disease activity in RA. The index was calculated using the following formula: CDAI: SJC28 + TJC28 + PGA (10 cm VAS) + PhGA (10 cm VAS + C-Reactive Protein (CRP). VAS assessments involved a 10-cm horizontal scale from 'no disease activity' to 'maximum disease activity. Scores ranged from 0 to 86, with higher scores also indicating increased disease activity.
Time Frame: Randomization (Week 24), Week 60, 72
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 136 | 136
percentage of participants
  Week 60 | 2.9 | 0.7
  Week 72 | 2.9 | 0.7

10. Secondary Outcome: Percentage of Participants With Improvement in Physical Function Using Health Assessment Questionnaire [HAQ] at Week 60 and 72
Description: The HAQ-disability index (DI) evaluates participant-reported quality of life using 8 categories: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and other common activities such as running errands and performing household chores and 20 questions. Each category contains multiple questions, which were answered using a 4-point scale from 0 to 3. The overall index score was an average of the individual item responses and may range from 0 to 3, where higher scores indicate more difficulty in daily living activities. Improvement was defined as a decrease from Week 24 to Week 60 and 72. Reported is the percentage of participants with an improvement in HAQ-DI score.
Time Frame: Randomization (Week 24), Week 60, 72
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 136 | 136
percentage of participants
  Improvement at Week 60 | 27.0 | 39.6
  Improvement at Week 72 | 40.5 | 50.0

11. Secondary Outcome: Percentage of Participants With Improvement in Physical Function Using Functional Assessment of Chronic Illness Therapy - Fatigue [FACIT-F] at Week 60 and 72
Description: The FACIT-fatigue assessment was a 13-item questionnaire with participants scoring each item on a 5-point scale (not at all; a little bit; somewhat; quite a bit and very much). The total score ranges from 0 to 65 and higher scores indicate more fatigue. Improvement was defined as a decrease from Week 24 to Week 60 and 72. Reported is the percentage of subjects with an improvement in total FACIT score.
Time Frame: Randomization (Week 24), Week 60, 72
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 136 | 136
percentage of participants
  Improvement at Week 60 | 54.0 | 50.0
  Improvement at Week 72 | 45.2 | 56.3

12. Secondary Outcome: Percentage of Participants With Improvement in Physical Function Using 12-item Short Form Health Survey [SF-12]) at Week 60 and 72
Description: Quality of life questionnaire (SF-12) scores were computed using the scores of 12 questions and ranged from 0 to 100, where a 0 score indicated the lowest level of health measured by the scales and 100 indicated the highest level of health. Improvement was defined as a decrease from Week 24 to Week 60 and 72. Reported is the percentage of subjects with an improvement in SF-12 score.
Time Frame: Randomization (Week 24), Week 60, 72
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 136 | 136
percentage of participants
  Improvement at Week 60 | 22.2 | 10.4
  Improvement at Week 72 | 23.8 | 15.6

13. Secondary Outcome: Percentage of Participants With Anemia
Time Frame: Week 0 up to Week 72
Population: Safety population included all the randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 136 | 136
percentage of participants | 1.5 | 0.7

14. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE was any adverse event that can be fatal, life threatening, requires long or prolong hospitalization, results in persistent or significant disability/incapacity, congenital anomaly or significant medical event in the investigator's judgment.
Time Frame: Week 0 up to Week 72
Population: Safety population included all the randomized participants.
Measure: Number; unit: participants
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 136 | 136
participants
  AEs | 98 | 98
  SAEs | 9 | 3

15. Secondary Outcome: Percentage of Participants Able to Discontinue Methotrexate
Time Frame: Week 0 up to Week 60
Population: Data were not collected for this outcome measure.
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Number of Subjects Employed Assessed Using the Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI-SHP)
Description: The WPAI-SHP questionnaire assesses work productivity and activity impairment. It is a patient-reported assessment regarding hours missed and hours worked at employment and degree to which a specified health problem affected work productivity and regular activities. It consists of 6 questions to assess the impact of a specific health problem on work productivity and on regular daily activities.
Time Frame: Randomization (Week 24), Week 60, 72
Population: ITT population included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 136 | 136
participants
  Week 60 | 33 | 17
  Week 72 | 23 | 14

17. Secondary Outcome: Hours Actually Worked and Work Hours Missed Assessed Using the WPAI-SHP
Description: The WPAI-SHP questionnaire assesses work productivity and activity impairment. It is a patient-reported assessment regarding hours missed and hours worked at employment and degree to which a specified health problem affected work productivity and regular activities. It consists of 6 questions to assess the impact of a specific health problem on work productivity and on regular daily activities. Reported here are hours actually worked, work hours missed due to rheumatoid arthritis (RA), work hours missed due to other reasons and the change from Week 24 for each of these parameters reported at Week 60 and Week 72.
Time Frame: Randomization (Week 24), Week 60, Week 72
Population: Participants in the ITT population with available data were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 136 | 136
hours
  Hours actually worked (HAW), Week 60 (n=33, 17) | 25.0 [0 to 58] | 28.0 [0 to 40]
  Change from Week 24 in HAW, Week 60 (n=29, 17) | -1.0 [-47 to 40] | 2.0 [-43 to 38]
  Work hours missed (WHM) to RA, Week 60 (n=33, 17) | 0.0 [0 to 15] | 0.0 [0 to 35]
  Change from Week 24 in WHM RA, Week 60 (n=30, 16) | 0.0 [-30 to 15] | 0.0 [-7 to 21]
  WHM other, Week 60 (n=33, 17) | 0.0 [0 to 46] | 0.0 [0 to 35]
  Change from Week 24 WHM other, Week 60 (n=30, 16) | 0.0 [-56 to 46] | 0.0 [-38 to 35]
  HAW, Week 72 (n=23, 13) | 30.0 [0 to 48] | 16.0 [0 to 40]
  Change from Week 24 in HAW, Week 72, (n=20, 12) | 0.0 [-37 to 23] | 2.5 [-30 to 40]
  WHM to RA, Week 72 (n=23, 13) | 0.0 [0 to 37] | 0.0 [0 to 35]
  Change from Week 24 in WHM RA, Week 72 (n=21, 11) | 0.0 [-30 to 37] | 0.0 [-7 to 21]
  WHM other, Week 72 (n=23, 13) | 0.0 [0 to 30] | 0.0 [0 to 8]
  Change from Week 24 WHM other, Week 72 (n=21, 11) | 0.0 [-56 to 30] | 0.0 [-38 to 2]

18. Secondary Outcome: Change in Productivity and Regular Daily Activities Affected by Rheumatoid Arthritis Assessed Using the WPAI-SHP
Description: The WPAI-SHP questionnaire assesses work productivity and activity impairment. It is a patient-reported assessment regarding hours missed and hours worked at employment and degree to which a specified health problem affected work productivity and regular activities. It consists of 6 questions to assess the impact of a specific health problem on work productivity and on regular daily activities. Assessments were made using a visual analogue scale ranging from 0 to 10 where 0 = minimum impact and 10 = maximum impact.
Time Frame: Randomization (Week 24), Week 60, 72
Population: Participants in the ITT population with available data at the respective time points were analyzed.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Number analyzed (Participants) | 136 | 136
units on a scale
  Productivity (P), Week 60 (n=34, 18) | 2.0 [0 to 8] | 2.0 [0 to 10]
  Change in P from Week 24 at Week 60 (n=30, 16) | 1.0 [-6 to 8] | 0.0 [-5 to 7]
  Regular Daily Activities (RDA), Week 60 (n=60, 45) | 3.0 [0 to 9] | 3.0 [0 to 9]
  Change in RDA from Week 24 at Week 60 (n=59, 44) | 0.0 [-5 to 7] | 0.0 [-6 to 6]
  Productivity (P), Week 72 (n=24, 12) | 3.0 [0 to 8] | 3.0 [0 to 9]
  Change in P from Week 24 at Week 72 (n=21, 11) | 0.0 [-3 to 4] | 0.0 [-5 to 7]
  Regular Daily Activities (RDA), Week 72 (n=42, 31) | 3.0 [0 to 10] | 3.0 [0 to 9]
  Change in RDA from Week 24 at Week 72 (n=41, 29) | 0.0 [-5 to 4] | -1.0 [-5 to 7]

ADVERSE EVENTS:
Time Frame: From start of treatment to unscheduled visit (up to Week 72)
Groups:
- Initial Phase: At Week 0 participants will start open-label tocilizumab and open-label MTX for 24 weeks, which is the initial phase of the study.
  Adverse events in this reporting group are those occurring in the open-label phase only.
- Methotrexate (MTX) Tapering Group: After the open-label period ended at Week 24, participants achieving a good/moderate European League Against Rheumatism (EULAR) disease response were randomized to the MTX Tapering Group or MTX Maintenance Group. In the MTX Tapering Group participants received a double-blind MTX dose according to the MTX tapering scheme between Week 24 and Week 56. In addition, participants continued to receive open-label tocilizumab between Week 24 and Week 56. From Week 56 to Week 72 participants received tocilizumab monotherapy.
  Adverse events in this reporting group are those occurring in the double-blind phase only.
- Methotrexate (MTX) Maintenance Group: After the open-label period ended at Week 24, participants achieving a good/moderate European League Against Rheumatism (EULAR) disease response were randomized to the MTX Tapering Group or MTX Maintenance Group. In the MTX Maintenance Group participants continued to be administered the same dose of MTX in a double-blind fashion from Week 25 to Week 56. In addition, participants continued to receive open-label tocilizumab from Week 25 to Week 56. From Week 56 to Week 72 participants received tocilizumab monotherapy.
  Adverse events in this reporting group are those occurring in the double-blind phase only.
Arm/Group | Initial Phase | Methotrexate (MTX) Tapering Group | Methotrexate (MTX) Maintenance Group
Serious Adverse Events (participants affected / at risk) | 21/427 | 9/136 | 3/136
Other Adverse Events (participants affected / at risk) | 263/427 | 62/136 | 70/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Phase (N=427) | Methotrexate (MTX) Tapering Group (N=136) | Methotrexate (MTX) Maintenance Group (N=136)
Diverticulitis (Infections and infestations) | 0 | 2 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 0
Abdominal Sepsis (Infections and infestations) | 0 | 1 | 0
Bursitis Infective (Infections and infestations) | 0 | 0 | 1
Lymph Node Tuberculosis (Infections and infestations) | 0 | 0 | 1
Necrotising Fasciitis (Infections and infestations) | 0 | 1 | 0
Device Dislocation (General disorders) | 0 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Arthritis Infective (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Clostridium Difficile Infection (Infections and infestations) | 1 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Tooth Infection (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Viral Labyrinthitis (Infections and infestations) | 1 | 0 | 0
Chest Pain (General disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Carcinoid Tumour Of The Gastrointestinal Tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Enterovesical Fistula (Gastrointestinal disorders) | 1 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 2 | 0 | 0
Blood Bilirubin Increased (Investigations) | 2 | 0 | 0
Carotid Artery Dissection (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Phase (N=427) | Methotrexate (MTX) Tapering Group (N=136) | Methotrexate (MTX) Maintenance Group (N=136)
Nasopharyngitis (Infections and infestations) | 61 | 16 | 17
Lower Respiratory Tract Infection (Infections and infestations) | 41 | 11 | 12
Upper Respiratory Tract Infection (Infections and infestations) | 23 | 12 | 7
Urinary Tract Infection (Infections and infestations) | 19 | 9 | 6
Diarrhoea (Gastrointestinal disorders) | 54 | 7 | 11
Mouth Ulceration (Gastrointestinal disorders) | 48 | 5 | 9
Nausea (Gastrointestinal disorders) | 28 | 5 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 8 | 9
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 13 | 7 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 16 | 2 | 7
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 23 | 9 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 8 | 6
Contusion (Injury, poisoning and procedural complications) | 16 | 7 | 6
Fall (Injury, poisoning and procedural complications) | 15 | 8 | 4
Headache (Nervous system disorders) | 38 | 8 | 6
Alanine Aminotransferase Increased (Investigations) | 51 | 6 | 7
Rash (Skin and subcutaneous tissue disorders) | 32 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.